CLINICAL TRIAL: NCT00057382
Title: T138067 Versus Doxorubicin in Chemotherapy-Naive, Unresectable, Hepatocellular Carcinoma Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tularik (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-067-010; NCT00066287 (obsolete NCT alias)
Record Dates: First submitted 2003-03-31; First posted 2003-04-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

INTERVENTIONS:
Drug: T138067 intravenous
Drug: doxorubicin intravenous

SUMMARY:
This is an international, multicenter, randomized study of intravenous T138067 versus intravenous doxorubicin in hepatocellular carcinoma (liver cancer). Patients can not have been treated before with chemotherapy and surgery is not recommended for their cancer. A total of 750 subjects will be enrolled in this study.

ELIGIBILITY:
Key inclusion criteria include:

* pathologic diagnosis of unresectable HCC
* chemotherapy-naïve for HCC
* Child-Pugh Class A or B liver disease
* measurable disease (i.e., at least one lesion that is at least 20 mm in one dimension) on computerized tomography (CT) scan or magnetic resonance imaging (MRI) or at least one lesion that is at least 10 mm on spiral CT scan
* Karnofsky Performance Status of ≥ 70%
* life expectancy of ≥ 12 weeks
* adequate hematologic function (i.e., absolute neutrophil count [ANC] of ≥ 1500 cells/mm3, platelet count of ≥ 80,000 cells/mm3, hemoglobin of ≥ 8.5 g/dL)
* total bilirubin of ≤ 1.5 upper limit of normal (ULN)
* aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 5 ULN
* serum creatinine of ≤ 2 x ULN

Key exclusion criteria include:

* severe, concurrent disease that would make the subject inappropriate for enrollment
* Subjects who have received prior intravenous or intra-arterial chemotherapy, chemoembolization, intratumoral ethanol injection, cryosurgery, radiofrequency ablation, or embolization for their HCC. (note: prior surgical resection, immunotherapy, hormonal therapy, radiotherapy, and/or orthotopic liver transplantation are allowed)
* history of other cancer within the past 5 years other than adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
* New York Heart Association (NYHA) class III or IV heart disease or a left ventricular ejection fraction of <50% or acute anginal symptoms
* females who are pregnant or breast-feeding
* received any investigational agent within 4 weeks of enrollment
* history of central nervous system metastases or carcinomatous meningitis
* clinically apparent ascites
* major surgery within 4 weeks of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hirmand, MD, Study Director — Tularik
Locations (76):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - University of California at San Francisco, San Francisco, California
  - VA Medical Center, Miami, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Loyola University of Chicago, Maywood, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center - Dallas, Dallas, Texas
- Brazil (4):
  - Hospital Vera Cruz, Belo Horizonte
  - Hospital Mater Dei - Departamento de Oncologia, Belo Horizonte
  - Irmandade Santa Casa de Misericórdia de Porto Alegre - Unidade de Apoio à Pesquisa, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo
- China (15):
  - Cancer Center, Sun Yat-Sen Unversity, Guangzhou, Guangdong
  - Guangzhou Nanfang Hospital, Guangzhou, Guangdong
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - Nanjing Ba Yi Hospital of PLA, Nanjing, Jiangsu
  - 1st Affiliated Hospital of Xi An Jiao Tong University, Xi’an, Shanxi
  - Taipei Veteran General Hospital, Taipei, Taiwan
  - Chang Gung Memorial Hospital, Taoyuan, Taiwan
  - Cancer Hospital of Chinese Academy of Medical Science (CAMS), Beijing
  - Beijing Cancer Hospital of Peking University, Beijing
  - Gereral Hospital of PLA, Beijing
  - Chongqing Southwest Hospital, Chongqing
  - Prince Wales Hosptial, Hong Kong
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Liver Cancer Institute, Zhongshan Hospital, Fudan University, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
- Poland (3):
  - Katedra i Klinika Onkologii i Radioterapi Akademii Medycznej, GdaDsk
  - Oddział Chemioterapii, Olsztyn
  - Klinika Katedry Onkologii AM, Poznan
- San Juan Medical Center, San Juan, Puerto Rico
- Russia (28):
  - Arkhangelsk Redional Oncology Center, Department of Chemotherapy, Arkhangelsk
  - Barnaul
  - Cheliabinsk Regional Oncology Center, Chelyabinsk
  - Irkutsk Regional Oncology Center, Irkutsk
  - Kazan State Medical University, Kazan'
  - Kazan Republican Oncology Clinical Center, Kazan'
  - Krasnodar City Oncology Center, Krasnodar
  - Krasnoyarsk Regional Oncology Center, Krasnoyarsk
  - Lipetsk, Lipetsk
  - Blokhin Cancer Research Center, Moscow
  - Central Clinical Hospital of the President of the Russian Federation, Moscow
  - Central Clinical Hospital of the Ministry of Transport, Moscow
  - Novosibirks Municipal Clinical Hospital #1, Novosibirsk
  - Russian Academy of Medical Sciences, Obninsk
  - Omsk Regional Oncology Center, Omsk
  - Orenburg Regional Oncology Center, Orenburg
  - Moscow Oncology Hospital #62, P/O Stepanovskoye
  - Rostov Research Oncology Institute, Rostov-on-Don
  - Central Research Institute of Radiology of the Ministry of Health of Russian Federation, Saint Petersburg
  - Medical Academy of Postgraduate Education, St. Petersburg, Saint Petersburg
  - St. Petersburg Mechnikov State Medical Academy, Saint Petersburg
  - St. Petersburg Oncology Center, Saint Petersburg
  - Stavropol Regional Oncology Center, Stavropol
  - Tomsk Regional Research Institute of Oncology, Tomsk
  - Bashkiria Republican Oncology Center, Ufa
  - Voronezh Regional Clinical Oncology Center, Voronezh
  - Yaroslavl Regional Oncology Center, Yaroslavl
  - Zhitomir Regional Hospital, Zhitomir
- National University Hospital, Singapore, Singapore
- Eastern Cape Oncology Centre, Port Elizabeth, South Africa
- Thailand (2):
  - Khon Kaen University, Khon Kaen
  - Chiangmai University, Muang Chiangmai
- Ukraine (9):
  - Dnepropetrovsk State Medical Academy, Dnipro
  - Donetsk Regional Antitumor Center, Donetsk
  - Kiev Central Military Clinical Hospital, Kiev
  - Kiev Oncology Institute of Ukrainian Academy of Medical Science, Kiev
  - Krivorojsky City Oncology Center, Kryvyi Rih
  - Lvov State Medical University, Lviv
  - Poltava Regional Clinical Oncological Center, Poltava
  - Vinnitsa Regional Clinical Oncological Center, Vinnitsa
  - Zaporozhje State Medical Institute of Postgraduate Education, Zaporizhzhya
- United Kingdom (4):
  - Addenbrookes Hospital, Cambridge
  - Royal Free Hospital, London
  - Hammersmith Hospital, London
  - Christie Hospital, Manchester